CLINICAL TRIAL: NCT07240428
Title: Comparison Between Interdental Brush and Water Floss on Plaque Accumulation and Gingival Inflammation in Patients Undergoing Fixed Orthodontic Treatment: A Single Blinded Split-Mouth Randomized Controlled Clinical Trial
Brief Title: Comparison Between Interdental Brush and Water Floss on Plaque Accumulation and Gingival Inflammation in Patients Undergoing Fixed Orthodontic Treatment.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Lana Bader, Dr, Assistant Professor, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 775/2023; 51/166/2024 (Other: Institutional Review Board at Jordan University of Science and Technology)
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Dental Plaque; Gingival Bleeding
Keywords: Interdental cleaning; Interdental brush; Water flosser; Oral hygiene; Orthodontic patients; Gingival inflammation; Plaque index; Oral irrigator
MeSH Terms: conditions — Dental Plaque; Gingival Hemorrhage; Gingivitis

STUDY DESIGN:
Intervention Model Description: Split-mouth randomized controlled clincal trial, where each participant receives one interdental cleaning method for the right side, and another one for the left side.
Who Masked: Investigator, Outcomes Assessor
Masking Description: patients know what they're using, but examiner measuring plaque/gingival index is blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interdental brush (Experimental): Participants used an interdental brush twice daily for interdental cleaning on the assigned side
  Interventions: Device: Interdental brush
- Water Flosser (Experimental): Participants used a water flosser twice daily for interdental cleaning on the other assigned side
  Interventions: Device: Water floss

INTERVENTIONS:
Device: Interdental brush — Participants used an interdental brush twice daily after toothbrushing on the assigned side. This method was compared to the use of water floss in the contralateral side (split-mouth design).
  Arms: Interdental brush
Device: Water floss — Participants used a water flosser twice daily after toothbrushing on the assigned side. Standard pressure setting and specialized tip were used. This method was compared to the use of an interdental brush in the contralateral quadrants (split-mouth design).
  Arms: Water Flosser

SUMMARY:
The goal of this clinical trial is to test the ability of water flosser to remove plaque and reduce gingival inflammation in patients undergoing fixed orthodontic treatment.

The main questions it aims to answer are:

Does water flosser remove plaque effectively in orthodontic patients? Does water flosser reduce gum inflammation in orthodontic patients?

Researchers compared water flosser to interdental brush to see if there is a difference in plaque and inflammation reduction.

Participants used interdental brush to clean between their teeth and around brackets in one side of their mouth, and they used water flosser to clean between the teeth and around brackets in the other side. The study lasted for 3 months.

DETAILED DESCRIPTION:
* Study design This is a randomized controlled single blinded clinical trial, with split mouth design.
* Sample size Forty seven subjects with fixed orthodontic appliance were recruited from patients attending dental teaching clinics at Jordan University of Science and Technology. The age range was between 18 and 35 years. They were randomly assigned to use interdental brush on one side of the mouth, and water floss on the other side in a split mouth design.

The study lasted for 3 months.

1. Inclusion criteria:

   1. Patients with fixed orthodontic appliance in the upper and lower arches. 2. Patients with healthy gingiva with no periodontal disease. 3. Patient's orthodontic plan doesn't require extraction of any teeth during the study period. .

   4. Patients should have at least 26 teeth. 5. Patients are motivated and able to clean their teeth. 6. Patients should not have caries, overhang restorations, crowns, bridges or implants 7. Adults 18-35 years old.
2. Exclusion criteria:

   1. Smokers 2. Medically compromised patients 3. Pregnant woman.
   * Ethical considerations The study was approved by the Institutional Review Board (IRB) of Jordan University of Science and Technology (51/166/2024). All participating patients were informed of the study's purpose, objectives, and methods. They all provided a written informed consent before data collection.
   * Data collection:

     1. Patients randomly used water floss on one side of the mouth , and the interdental brush on the other side.
     2. Randomization was used to assign the intervention to either the left or right side of the mouth.

        The following will be assessed

        1- Plaque score using Rustogi modified navy plaque index for buccal and lingual surfaces, where the tooth was divided into multiple zones as the following :

        The divided zones are:

        Whole mouth: areas A,B,C,D,E,F,G and H. Marginal (gum line): areas A,B and C. Interproximal: areas D and F

        0 score was given the area where there is no plaque.

        1 score was given in the area where there is plaque Intraoral photos using professional camera were taken for all teeth and all surfaces to record the plaque score.

        2. gingival inflammation was recorded using gingival index at six sites per tooth (distobuccal, midbuccal, mesiobuccal, distolingual/palatal, midlingual/palatal, mesiolingual/palatal) as follows : 0= Normal gingiva.
        1. Mild inflammation - slight change in colour and slight edema but no bleeding on probing.
        2. Moderate inflammation - redness, edema and glazing, bleeding on probing.
        3. Severe inflammation - marked redness and edema, ulceration with tendency for spontaneous bleeding.

        3.Visual Analog Scale (VAS) visual analog scale from 0 - 10 (0 - unsatisfied, uncomfortable, or difficult to use, 10 -very satisfied, comfortable, and easy to use) in each visit was taken.

        Randomization and Blinding Independent of the clinical assessment, a third-party dentist used a computer-generated random number sequence to determine which side of each patient's mouth will be cleaned by interdental brush and which side will be cleaned by the oral irrigator. While participants were aware of which device they were using on each side, the examiner who performed the clinical examinations was blinded.
   * Adverse events monitoring: Participants were monitored for adverse events during the study period such as gingival trauma, sensitivity, recession, tooth or restoration damage.

ELIGIBILITY:
Inclusion Criteria:

* Patients with fixed orthodontic appliance upper and lower arches.
* Patients with healthy gingiva with no periodontal disease.
* Patient's orthodontic plan doesn't require extraction of any teeth during the study period.
* Patients should have at least 26 teeth.
* Patients are motivated and able to clean their teeth.
* Patients should not have caries, overhang restorations, crowns, bridges or implants.
* Adults 18-35 years old.

Exclusion Criteria:

* Smokers.
* Medically compromised patients.
* Pregnant woman.
* Using mouth wash or antibiotic in last 3 months.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Plaque Index | Baseline, 2 weeks, 4 weeks, 2 month and 3 months
  Plaque accumulation assessed using the Rustogi Modified Navy Plaque Index (RMNPI) on designated tooth surfaces in the sides assigned to interdental brush and water flosser. The tooth was divided into multiple zones as the following :
  Whole mouth: areas A,B,C,D,E,F,G and H. Marginal (gum line): areas A,B and C. Interproximal: areas D and F
  0 score was given the area where there is no plaque.
  1 score was given in the area where there is plaque The minimum plaque score per surface (buccal or lingual) is zero, and the maximum plaque score per surface is 8 Intraoral photos using professional camera were taken for all teeth and all surfaces to record the plaque score.

SECONDARY OUTCOMES:
Gingival Index | Baseline, 2 weeks, 4 weeks, 2 months ,and 3 months
  Gingival inflammation was recorded using gingival index at six sites per tooth (distobuccal, midbuccal, mesiobuccal, distolingual/palatal, midlingual/palatal, mesiolingual/palatal) in each intervention side as follows :
  0= Normal gingiva.
  1. Mild inflammation - slight change in colour and slight edema but no bleeding on probing.
  2. Moderate inflammation - redness, edema and glazing, bleeding on probing.
  3. Severe inflammation - marked redness and edema, ulceration with tendency for spontaneous bleeding.
  The minumn score is zero and the maximum score for one surface (buccal or lingual/palatal is 9.
Visual Analog Scale (VAS) | 2 Weeks, 4 weeks, 2months, and 3months
  visual analog scale from 0 - 10 (0 - unsatisfied, uncomfortable, or difficult to use, 10 -very satisfied, comfortable, and easy to use)

CONTACTS AND LOCATIONS:
Overall Officials: Lana Bader, DClinDent, Study Director — Jordan University of Science and Technology; Reem Sami Abed Alhafez, DClinDent Perio, Study Director — Jordan University of Science and Technology; Ahmad shawqi, MClinDent Perio, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and Technology, Faculty of Dentistry, Irbid, Irbid Governorate, Jordan

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data for plaque index (RMNPI), gingival index and patient-reported outcomes will be shared. Data will be stripped of all identifiers to protect participants privacy.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD and supporting documents will be available after publication of the main study results, for a period of one year.
Access Criteria: Access will be granted to qualified researchers who request the data via email to the principal investigator. Researchers must sign a data use agreement ensuring ethical use, confidentiality, and prohibition of attempts to identify participants.